CLINICAL TRIAL: NCT06076837
Title: An Open-label, Phase I Trial With Expansion Cohort of Nab-Paclitaxel + Gemcitabine + Cisplatin + Botensilimab (AGEN1811) + Balsilimab (AGEN2034) + Chloroquine + Celecoxib in Patients With Previously Untreated Metastatic Pancreatic Cancer
Brief Title: The Seven Trial: Exploiting the Unfolded Protein Response
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Collaborators: University of Arizona (Other); Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HRI-2023 Magnificent 7
Record Dates: First submitted 2023-09-21; First posted 2023-10-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer Metastatic; Pancreatic Adenocarcinoma Metastatic
MeSH Terms: interventions — balstilimab; chloroquine diphosphate; Chloroquine; Celecoxib; Taxes; Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: (Part 1) Maximum Tolerated Dose (MTD) Safety Group; (Part 2) Expansion Cohort - Botensilimab MTD from Part 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DoseEscalationBotensilimab+balstilimab+nab-paclitaxel+gemcitabine+cisplatin +chloroquine + celecoxib (Experimental): Botensilimab 50 mg IV, Balstilimab 240 mg, nab-paclitaxel 125 mg/m2 + gemcitabine 1000 mg/m2 +cisplatin 25 mg/m2; Chloroquine phosphate 500 mg po (300 mg equivalent chloroquine base); Celecoxib 200 mg po twice daily (BID) on Famotidine 20 mg po BID Aspirin 81 mg
  Interventions: Drug: Botensilimab; Drug: Balstilimab; Drug: Chloroquine Phosphate; Drug: Celecoxib; Drug: Nab paclitaxel; Drug: Gemcitabine; Drug: Cisplatin
- Expansion Cohort-Botensilimab+balstilimab+nab-paclitaxel+gemcitabine+cisplatin+chloroquine+celecoxib (Experimental): Botensilimab (MTD TBD), Balstilimab 240 mg IV, nab-paclitaxel 125 mg/m2 + gemcitabine 1000 mg/m2 +cisplatin 25 mg/m2 IV infusion ; Chloroquine phosphate 500 mg po (300 mg equivalent chloroquine base),Celecoxib 200 mg po twice daily (BID); Famotidine 20 mg po BID Aspirin 81 mg
  Interventions: Drug: Botensilimab; Drug: Balstilimab; Drug: Chloroquine Phosphate; Drug: Celecoxib; Drug: Nab paclitaxel; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Botensilimab — an Fc-engineered anti-CTLA-4 (cytotoxic T-lymphocyte antigen 4) monoclonal antibody
  Other Names: AGEN1811
Drug: Balstilimab — a human monoclonal immunoglobulin (Ig) G4 (IgG4) antibody, designed to block programmed cell death protein (PD-1) binding by PD-L1 and PD-L2
  Other Names: AGEN2034
Drug: Chloroquine Phosphate — an antimalarial agent, that is being used in this patient population to sensitize cancer cells to chemotherapy and leads to anticancer effects through inhibiting autophagy
  Other Names: Aralen
Drug: Celecoxib — a second-generation selective Cyclooxygenase 2 (COX-2) inhibitor, is being used in this patient population to enhance the therapeutic effect of cisplatin by inhibiting the expression of COX-2 as well as inhibit anti-apoptotic gene BCL-2 (B-cell lymphoma 2)
  Other Names: Celebrex
Drug: Nab paclitaxel — microtubule inhibitor indicated for the treatment of Metastatic adenocarcinoma of the pancreas as first-line treatment, in combination with gemcitabine
Drug: Gemcitabine — a nucleoside metabolic inhibitor indicated as a single agent for the treatment of pancreatic cancer
Drug: Cisplatin — platinum-based drug indicated for the treatment of advanced cancers

SUMMARY:
The goal of this investigator initiated interventional study is to improve the response to the anticancer treatments (chemotherapy) in people who have previously untreated metastatic pancreas cancer. The main question it aims to answer is:

• Do new types of immune-based therapies, called botensilimab, and balstilimab, when given in combination with chemotherapy consisting of nab-paclitaxel + gemcitabine + cisplatin, and oral medications of chloroquine and celecoxib help patients with previously untreated metastatic pancreatic cancer?

Participants will be administered two immune-based therapies:

* Botensilimab (also referred to as AGEN1811)
* Balstilimab (also referred to as AGEN2034)

Patients will be evaluated when given in combination with:

* Triple chemotherapy (nab-paclitaxel + gemcitabine + cisplatin), plus two oral medications:
* chloroquine
* celecoxib

DETAILED DESCRIPTION:
This Investigator Initiated Trial (IIT) is proposed based on our experience of obtaining high response rates with chemotherapy or chemotherapy + Programmed cell death protein 1 (PD1) checkpoint inhibitor in patients with previously untreated stage 4 pancreatic adenocarcinoma. However, investigators have hit a barrier as they have not been able to improve the complete response rate above 20% nor improve the 64% 2-year survival rate. For the most part ultimately, the patient's tumor progresses.

Pancreatic cancer relies upon unfolded protein response (UPR) to for survival. The endoplasmic reticulum has stress stressors with a variety of proteins that when activated during stress promote proteostasis and homeostasis which prevents apoptosis. While the UPR is able to achieve homeostasis, under prolonged and unresolved stress, the signaling pathway will lead to apoptosis. In pancreatic cancer, the UPR does play a role as it is upregulated to allow for greater survival. Prior cancer research has been focused on mitigating UPR in cancer through agents such as HSP90 inhibitors but this has not been successful. The hypothesis of this study is that by increasing ER stress and thus UPR that apoptosis occurs in pancreatic cancer by the use of these agents and improve the survival in individuals with advanced pancreatic cancer.

Visually it looks like this with three possibilities when tumor cells are under stress:

1. They survive
2. They go into dormancy
3. They undergo apoptosis

Investigators seek to increase ER stress (UPR) to drive that system to apoptosis. To achieve the apoptosis, the investigators seek the maximum treatment approach with maximum chemo immunotherapy to stress the tumor cells (increase of ER stress /UPR) and use 2 agents to help block escape routes a) block autophagy via chloroquine and b) block microenvironment inflammation via celecoxib.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate by giving signed, dated, and written informed consent prior to any study-specific procedures.
2. ≥ 18 years of age.
3. Histologically confirmed diagnosis of metastatic pancreatic ductal adenocarcinoma.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix A).
5. Life expectancy of at least 3 months.
6. Measurable disease on baseline imaging per RECIST 1.1 criteria.
7. < Grade 2 pre-existing peripheral neuropathy per NCI CTCAE, Version 5.0.
8. Acceptable coagulation status as indicated by an international normalized ratio (INR)

   * 1.5 times institutional upper limit of normal (ULN), except patients on anticoagulation who can be included at the discretion of the investigator.
9. Adequate organ function defined as the following laboratory values within 7 days prior to first dose of study drugs, except where noted below:

   1. Neutrophils > 1500/μL (stable off any growth factor within 4 weeks prior to first dose of study drugs).
   2. Platelets > 100 × 103/μL (transfusion to achieve this level is not permitted within 2 weeks prior to first dose of study drugs).
   3. Hemoglobin > 9.0 g/dL (transfusion to achieve this level is not permitted within 2 weeks prior to first dose of study drugs).
   4. Creatinine of < 1.5mg/dL or Creatinine clearance ≥ 45 mL/min (measured or calculated per institutional standards).
   5. Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) < 3.0 × ULN.
   6. Total bilirubin < 1.25 × ULN (except patients with Gilbert syndrome who must have a total bilirubin level of < 3.0 × ULN).
   7. Serum albumin ≥ 3.0 g/dL (must be confirmed within 3 days prior to first dose of study drugs).
10. Female patients of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test at screening (within 72 hours of first dose of study drugs).

    WOCBP must agree to use highly effective contraceptive measures starting with the screening visit through 6 months after the last dose of study drug(s). Highly effective contraception is defined in Appendix B, Guidance on Contraception, or as stipulated in national or local guidelines. Non-childbearing potential is defined as:
    1. ≥ 50 years of age and has not had menses for greater than 1 year.
    2. Amenorrheic for ≥ 2 years without a hysterectomy and/or bilateral oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre- study (screening) evaluation.
    3. Status is post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation.
11. Male patients with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the study starting with the screening visit through 6 months after the last dose of study drug(s) is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.
12. Willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Patients must have received no previous radiotherapy, surgery, chemotherapy, or investigational therapy for the treatment of metastatic disease. Prior treatments in the adjuvant setting with gemcitabine and/or 5-Fluorouracil (5-FU) or gemcitabine administered as a radiation sensitizer are allowed, provided at least 6 months have elapsed since completion of the last dose and development of metastatic disease and no lingering toxicities are present.
2. History of central nervous system (CNS) metastasis.
3. Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to the first dose of study drugs (i.e., patients with a history of prior malignancy are eligible if treatment was completed at least 2 years prior to first dose of study drugs and the patient has no evidence of disease). Patients with history of prior early-stage basal/squamous cell skin cancer or noninvasive or in situ cancers who have undergone definitive treatment at any time are also eligible.
4. QTc Derived From Fridericia's Formula (QTcf) > 450 ms on electrocardiogram (ECG)
5. Uncontrolled intercurrent illness, including but not limited to clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ III), or serious uncontrolled cardiac arrhythmia requiring medication. Patients with history of coronary bypass procedure are ineligible.
6. Active, uncontrolled infections, requiring systemic intravenous anti-infective treatment within 2 weeks prior to first dose of study drugs.
7. Major surgery within 4 weeks prior to signing of informed consent form (ICF).
8. Prior treatment with an immune checkpoint inhibitor.
9. Refractory ascites defined as requiring 2 or more therapeutic paracenteses within the last 4 weeks or ≥ 4 within the last 90 days or ≥ 1 time within the last 2 weeks prior to signing of ICF or requiring diuretics intended to treat ascites within 2 weeks of signing of ICF.
10. Partial or complete bowel obstruction within the last 3 months prior to signing of ICF, signs/symptoms of bowel obstruction, or known radiologic evidence of impending obstruction.
11. Clinically significant gastrointestinal (GI) disorders including:

    1. GI perforation or unhealed ulcerations < 6 months prior to signing of ICF. Patients must have documented evidence (e.g., upper endoscopy, colonoscopy) of completely healed area of prior perforation or ulceration.
    2. Clinically significant GI bleeding < 3 months prior to signing of informed consent.
    3. History of active Crohn's disease or ulcerative colitis.
12. Previous severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to first dose of study drugs.
13. SARS-CoV-2 vaccine < 7 days prior to first dose of study drugs.
14. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
15. Symptomatic interstitial lung disease (ILD), history of ILD, or any lung disease which may interfere with detection and management of new immune-related pulmonary t toxicity.
16. History of allogeneic organ transplant.
17. Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
18. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) within 14 days or another immunosuppressive medication within 30 days prior to the first dose of study drugs. Inhaled or topical steroids, and adrenal replacement steroid doses (≤ 10 mg daily prednisone equivalent), are permitted in the absence of active autoimmune disease.
19. Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years prior to first dose of study drugs (i.e., with use of disease- modifying agents or immunosuppressive drugs).
20. Pregnant or breastfeeding patients.
21. Uncontrolled infection with HIV. Patients on stable highly active antiretroviral therapy ( (HAART) therapy with undetectable viral load and normal CD4 (Cluster of differentiation 4) counts for at least 6 months prior to signing ICF. Serological testing for HIV at screening is to be performed at the investigator's discretion based on individual patient's risk factors.
22. Known to be positive for hepatitis B (HBV) surface antigen, or any other positive test for HBV indicating acute or chronic infection. Patients who are or have received anti-HBV therapy are eligible, permitting they have undetectable HBV DNA for at least 6 months prior to signing ICF. Serological testing for HBV at screening is to be performed at the investigator's discretion based on the individual patient's risk factors.
23. Known active hepatitis C (HCV) as determined by positive serology and confirmed by polymerase chain reaction (PCR). Patients on or having received antiretroviral therapy are eligible provided they are virus-free by PCR for at least 6 months prior to signing ICF. Serological testing for HCV at screening is to be performed at the investigator's discretion based on individual patient's risk factors.
24. Dependence on total parenteral nutrition.
25. Patients with concurrent diarrhea > grade 1 at time of enrollment despite optimal treatment with standard of care pancreatic enzymes.
26. Known active or latent tuberculosis (testing at screening not required).
27. Any condition in the opinion of the principal investigator that might interfere with the patient's participation in the study or in the evaluation of the study results.
28. Unwillingness or inability to comply with procedures required in this protocol.
29. History of coronary artery bypass graft.
30. Patients receiving warfarin or digoxin.
31. Presence of retinal or visual field changes of any etiology. Note: An ophthalmological examination to be performed within the 3 weeks of starting Chloroquine (C1/D1) to include: best corrected distance visual acuity (BCVA), an automated threshold visual field (VF) of the central 10 degrees (with retesting if an abnormality is noted), and spectral domain optical coherence tomography (SD-OCT). All of these parameters should be within normal parameters.
32. Known hypersensitivity to 4-aminoquinoline compounds (chloroquine, hydroxychloroquine, and amodiaquine).
33. Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
34. History of asthma, urticaria, or other allergic-type reactions after taking aspirin or other NSAIDs.
35. Patients who have demonstrated allergic-type reactions to sulfonamides.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 12 months
  To determine the maximum tolerated dose (MTD) of botensilimab when given in combination with balstilimab + triplet chemotherapy regimen (consisting of nab-paclitaxel + gemcitabine + cisplatin) + chloroquine + celecoxib to be used in Part 2-Dose Expansion. MTD will be defined at the dose of botensilimab at which no more than 1 of 6 evaluable patients experiences a dose-limiting toxicity (DLT).
Safety and Tolerability of botensilimab in combination with balstilimab + triplet + chloroquine + celecoxib. Treatment-related toxicities as per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTC AE V5.0). | End of Study (up to 2 years)
  To evaluate the safety and tolerability of botensilimab in combination with balstilimab + triplet + chloroquine + celecoxib. Treatment-related toxicities as per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTC AE V5.0).

SECONDARY OUTCOMES:
Complete Response (CR) | End of Study (up to 2 years)
  To determine the preliminary efficacy of botensilimab at the MTD + balstilimab + triplet + chloroquine + celecoxib in patients with previously untreated metastatic pancreatic cancer. Complete Response (CR) rate as defined by CT scan using RECIST 1.1 criteria, the overall response rate (ORR), progression free survival (PFS) and overall survival (OS).
Overall Response Rate (ORR) | End of Study (up to 2 years)
  To determine the preliminary efficacy of botensilimab at the MTD + balstilimab + triplet + chloroquine + celecoxib in patients with previously untreated metastatic pancreatic cancer. Complete Response (CR) rate as defined by CT scan using RECIST 1.1 criteria, the overall response rate (ORR), progression free survival (PFS) and overall survival (OS).
Progression free survival (PFS) | End of Study (up to 2 years)
  To determine the preliminary efficacy of botensilimab at the MTD + balstilimab + triplet + chloroquine + celecoxib in patients with previously untreated metastatic pancreatic cancer. Complete Response (CR) rate as defined by CT scan using RECIST 1.1 criteria, the overall response rate (ORR), progression free survival (PFS) and overall survival (OS).
Overall Survival (OS) | End of Study (up to 2 years)
  To determine the preliminary efficacy of botensilimab at the MTD + balstilimab + triplet + chloroquine + celecoxib in patients with previously untreated metastatic pancreatic cancer. Complete Response (CR) rate as defined by CT scan using RECIST 1.1 criteria, the overall response rate (ORR), progression free survival (PFS) and overall survival (OS).
Disease Control Rate (CR), Partial Response (PR), and Stable Disease (SD) | 12 Weeks
  To evaluate the disease control rate (CR, PR, and SD at 12 weeks) at the MTD of botensilimab + balstilimab + triplet + chloroquine + celecoxib in patients with previously untreated metastatic pancreatic cancer. Disease control rate (CR, PR, and SD at 12 weeks) using RECIST 1.1 criteria.
CA 19-9 (or CA 125, or CEA if not expressers of CA 19-9) | End of Study (up to 2 years)
  To evaluate the change in carbohydrate antigen 19-9 (CA 19-9) (or cancer antigen 125 [CA 125], or carcinoembryonic antigen [CEA] if not expressers of CA 19-9) in this patient population. Change from start of treatment CA 19-9 (or CA 125, or CEA if not expressers of CA 19-9).
  Rates of normalization of CA 19-9 (or CA 125, or CEA if not expressers of CA 19-9).

OTHER OUTCOMES:
Quality of Life: MD Anderson Symptom Inventory (MDASI-GI) | through study completion (up to 3 years)
  To evaluate the participant's self-reported quality of life during this study. Participant's self-reported quality of life and pain levels during this study utilizing the MD Anderson Symptom Inventory (MDASI-GI). This questionnaire asks about severity of symptoms using numbers (0 = not present to 10 = as bad as you can imagine).
Pain Levels: Brief Pain Inventory (BPI) | through study completion (up to 3 years)
  To evaluate the participant's self-reported pain levels during this study. Participant's self-reported quality of life and pain levels during this study utilizing the Brief Pain Inventory (BPI). This form asks about severity of pain using numbers (0 = not present to 10 = as bad as you can imagine).
Determination of the Effects of the regimen - ER stress (unfolded protein response) level assessment | through study completion (up to 3 years)
  Doubling of levels (over baseline) of 78 KDa Glucose regulated protein (GRP78) stress response marker in plasma.
Determination of the Effects of the regimen - Molecular Response assessment | through study completion (up to 3 years)
  Measuring the decrease in circulating tumor deoxyribonucleic acid (ctDNA) mutational markers in patients who become minimal residual disease (MRD) negative.
Baseline neutrophil lymphocyte ratio (NLR) | through study completion (up to 3 years)
  To compare the survival rates based on baseline neutrophil lymphocyte ratio (NLR). NLR ≤5 versus NLR >5.
  Survival is defined as the time from enrollment to date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Nurse Navigator, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malhotra JD, Kaufman RJ. The endoplasmic reticulum and the unfolded protein response. Semin Cell Dev Biol. 2007 Dec;18(6):716-31. doi: 10.1016/j.semcdb.2007.09.003. Epub 2007 Sep 8. PMID 18023214
- [Background] Botrus G, Miller RM, Uson Junior PLS, Kannan G, Han H, Von Hoff DD. Increasing Stress to Induce Apoptosis in Pancreatic Cancer via the Unfolded Protein Response (UPR). Int J Mol Sci. 2022 Dec 29;24(1):577. doi: 10.3390/ijms24010577. PMID 36614019